CLINICAL TRIAL: NCT06601231
Title: Addition of GAAD Score to Imaging Surveillance for Early Identification of Liver Cancer.
Brief Title: To Quantify the Impact of Addition of the GAAD Score to Imaging in Patients with Chronic Liver Disease Eligible for HCC Surveillance.
Acronym: ADRENALIN
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Milan Sonneveld, Associate Professor, Erasmus Medical Center
Other Study IDs: NL85202.078.23
Record Dates: First submitted 2024-04-22; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer, Hepatocellular
Keywords: GAAD score; early detection
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample material is obtained during regular blood assessment. For the purpose of biobanking, a maximum of 20mL of additional blood will be drawn and stored in for future studies. The central biobank has given approval for the storage of the samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all patients who are eligible for HCC surveillance: All patients with cirrhosis
  * Non-cirrhotic chronic hepatitis B patients meeting any of the following criteria: positive family history for HCC, intermediate-high aMAP and/or (m)PAGE-B score (if non-Caucasian)
  * Non-cirrhotic chronic hepatitis C patients (with or without SVR) with a history of F3 fibrosis (based on histology or liver stiffness assessment)
  * Non-cirrhotic NASH patients with a history of F3 fibrosis (based on histology or liver stiffness assessment)
  Interventions: Diagnostic Test: GAAD score

INTERVENTIONS:
Diagnostic Test: GAAD score — In order to calculate the GAAD score an in-vitro diagnostic is used. The Elecsys GAAD assay by Roche Diagnostics is used to assess the GAAD score using on blood samples collected from patients during regular outpatient clinic visits. The Elecsys GAAD test combines the results of the Elecsys PIVKA-II and Elecsys AFP assays with gender and age (the GAAD score is calculated with PIVKA-II, AFP, gender and age).

SUMMARY:
The goal of this prospective observational study is to test the impact of addition of the GAAD score to imaging in patients with chronic liver disease eligible for HCC surveillance. The main questions it aims to answer are:

* Diagnostic accuracy of the GAAD score (cut-off 2.57 (3)) for detection of HCC (overall and by BCLC stage), expressed using sensitivity, specificity, negative predictive value and positive predictive value.
* Change in GAAD score over time, and proportion of patients with a GAAD score above the cut-off over time in relation to potential confounding factors (e.g. age, bilirubin levels, presence of HCC).

  1000 participants with chronic liver disease eligible for HCC surveillance will be enrolled. Data will be collected for 3 consecutive years after enrollment. As per clinical practice, patients will undergo standard bi-annual HCC surveillance comprising liver imaging with ultrasound (or CT or MRI based on previous investigations) and GAAD score assessment based on blood samples.

ELIGIBILITY:
Inclusion Criteria:

* All patients with cirrhosis
* Non-cirrhotic chronic hepatitis B patients meeting any of the following criteria: positive family history for HCC, intermediate-high aMAP and/or (m)PAGE-B score (if non-Caucasian)
* Non-cirrhotic chronic hepatitis C patients (with or without SVR) with a history of F3 fibrosis (based on histology or liver stiffness assessment)
* Non-cirrhotic NASH patients with a history of F3 fibrosis (based on histology or liver stiffness assessment)

Exclusion Criteria:

* Diagnosis with any other cancer other than non-melanoma skin cancer
* History of HCC
* Women who are pregnant or lactating
* Patient with glomerular filtration rate <45 ml /min/1.73 m2
* Unwillingness or inability to undergo both CT and MRI imaging
* Life expectancy <2 years
* Use of vitamin K antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (18 years or older) patients with chronic liver disease, with an indication for HCC surveillance, are potentially eligible for enrolment.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value of the GAAD score for HCC | 6 months
  The diagnostic value of the GAAD score for HCC will be expressed using sensitivity, specificity, positive and negative predictive values, both overall and for the subgroup of early stage (BCLC 0-A) HCC. The GAAD scores will be measured and documented separately for each visit. The diagnostic value of the GAAD score will be assessed for HCC diagnosed at the index visit (ie the visit at which the GAAD score was determined) and for HCC diagnosed on imaging performed at 6 months after the index visit.

SECONDARY OUTCOMES:
Change in GAAD score over time in relation to confounding factors | 3 years
  Change in GAAD score over time in relation to confounding factors will be analysed using pairwise comparisons and linear regression. The following confounding factors will be analysed: age in years, gender, ALT, creatinine umol/L and bilirubin U/L. The proportion of patients with a GAAD score above the cut-off will be shown using descriptive statistics. The association between the occurrence of HCC in relation to the change in GAAD score, (from below to above the cut-off score) will be expressed using sensitivity, specificity, positive and negative predictive values as described above.

CONTACTS AND LOCATIONS:
Overall Officials: M. J. Sonneveld, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, CA, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Yang JD, Addissie BD, Mara KC, Harmsen WS, Dai J, Zhang N, Wongjarupong N, Ali HM, Ali HA, Hassan FA, Lavu S, Cvinar JL, Giama NH, Moser CD, Miyabe K, Allotey LK, Algeciras-Schimnich A, Theobald JP, Ward MM, Nguyen MH, Befeler AS, Reddy KR, Schwartz M, Harnois DM, Yamada H, Srivastava S, Rinaudo JA, Gores GJ, Feng Z, Marrero JA, Roberts LR. GALAD Score for Hepatocellular Carcinoma Detection in Comparison with Liver Ultrasound and Proposal of GALADUS Score. Cancer Epidemiol Biomarkers Prev. 2019 Mar;28(3):531-538. doi: 10.1158/1055-9965.EPI-18-0281. Epub 2018 Nov 21. PMID 30464023
- [Background] Piratvisuth T, Hou J, Tanwandee T, Berg T, Vogel A, Trojan J, De Toni EN, Kudo M, Eiblmaier A, Klein HG, Hegel JK, Madin K, Kroeniger K, Sharma A, Chan HLY. Development and clinical validation of a novel algorithmic score (GAAD) for detecting HCC in prospective cohort studies. Hepatol Commun. 2023 Nov 8;7(11):e0317. doi: 10.1097/HC9.0000000000000317. eCollection 2023 Nov 1. PMID 37938100
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764